CLINICAL TRIAL: NCT05080790
Title: Combined Treatment With Dinutuximab Beta, Zoledronic Acid and Low-dose Interleukin (IL-2) in Patients With Metastatic or Inoperable Leiomyosarcoma - DiTuSarc Study
Brief Title: Treatment With Dinutuximab Beta, Zoledronic Acid and Low-dose Interleukin (IL-2) in Patients With Leiomyosarcoma
Acronym: DiTuSarc
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Collaborators: RECORDATI GROUP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DiTuSarc / GISG-20
Record Dates: First submitted 2021-07-15; First posted 2021-10-18 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Leiomyosarcoma
MeSH Terms: conditions — Leiomyosarcoma | interventions — dinutuximab; Zoledronic Acid; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 5 cycles (Q5W) of dinutuximab beta, interleukin-2 and zoledronic acid (Experimental): 5 cycles (Q5W) of dinutuximab beta, 20mg/m2/day, interleukin-2, 5.4x10^6, and zoledronic acid, 4 mg
  Interventions: Drug: Dinutuximab Beta, Zoledronic acid, Interleukin-2

INTERVENTIONS:
Drug: Dinutuximab Beta, Zoledronic acid, Interleukin-2 — Five 5-week cycles (Q5W) of dinutuximab beta, zoledronic acid and low-dose interleukin (IL-2)

SUMMARY:
Dinutuximab beta was designed to bind to neuroblastoma cells and other cancer cells that express the GD2 antigen, such as STS/LMS cells, and it is believed that this binding "labels" the cells an makes them a better target.

In addition, γδ T cells can safely be expanded in-vivo using intravenous zoledronic acid and subcutaneous interleukin-2 (IL-2) in patients with different types of solid tumors [Dieli et al., 2007; Pressey et al., 2016].

It is supposed that combination treatment using dinutuximab beta, zoledronic acid and IL-2 is more effective than their use in isolation. The already-established safety profiles of these agents make testing of the combination in GD2 positive cancers such as GD2 expressing LMS both rational and feasible [Fisher et al., 2015].

DETAILED DESCRIPTION:
Soft-tissue sarcomas (STS) are a heterogeneous group of malignancies characterized by both their relatively low incidence and their poor prognosis, encompassing more than 60 distinct diagnoses. Leiomyosarcoma (LMS), together with liposarcoma, is one of the most frequent sub-types amongst STS and accounts for up to 25% of all newly diagnosed STS [Guo et al., 2015].

The absence of definite causative risk factors for LMS, whether genetic, epigenetic or environmental, make this disease particularly difficult to understand and difficult to treat.

Classically, soft-tissue sarcomas (STS) have been treated as a single disease and with LMS as one of the most frequent sub-types the results with conventional therapies have been rather disappointing, especially in the advanced setting. The use of novel therapeutic approach such immunotherapy has also not yielded the same success compared to other tumor entities, whereas the heterogeneity of this malignancy certainly plays a role.

Current immunotherapy trials mostly use monoclonal antibodies to target those molecules or interactions, that essentially "take the brakes off" the immune system. If the underlying immune response however is poor, simply taking the brakes off will be insufficient. In tumors that do not trigger a sufficient immune response, it might be an advantages strategy to try make the tumor a better target and thus trigger a better antitumor immune response.

Strategies that incorporate the tumoricidal properties of gammadelta T cells (γδ T cells) represent a promising immunotherapeutic strategy for treatment of solid malignancies including neuroblastoma (NB) [Dieli et al., 2007]. An evaluation of pooled data from 132 published in vitro experiments shows a consistent improvement in the cytotoxicity of γδ T cells in the presence of antitumor antibodies. Immunotherapy using γδ T cells alone shows promising clinical activity, but there is a strong preclinical rationale for combining this treatment modality with cancer-targeting antibodies to augment its efficacy [Fisher et al., 2014].

Dinutuximab beta was designed to bind to neuroblastoma cells and other cancer cells that express the GD2 antigen, such as STS/LMS cells, and it is believed that this binding "labels" the cells an makes them a better target.

In addition, γδ T cells can safely be expanded in-vivo using intravenous zoledronic acid and subcutaneous interleukin-2 (IL-2) in patients with different types of solid tumors [Dieli et al., 2007; Pressey et al., 2016].

It is supposed that combination treatment using dinutuximab beta, zoledronic acid and IL-2 is more effective than their use in isolation. The already-established safety profiles of these agents make testing of the combination in GD2 positive cancers such as GD2 expressing LMS both rational and feasible [Fisher et al., 2015].

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed leiomyosarcoma.
2. ≥ 1 prior systemic therapy for sarcoma, including adjuvant systemic therapy (anthracycline-containing regimen).
3. Patients must have a cryopreserved and formalin-fixed paraffin-embedded tumor sample available for submission to central pathology review.
4. Signed Written Informed Consent.
5. Men and women aged ≥ 18 years.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
7. Measurable disease.
8. Locally advanced/unresectable or metastatic disease.
9. No prior therapy with any agent targeting GD2.
10. Confirmed GD2-Expression proven on cryopreserved tissue tumor samples. A staining score of 2 on cryopreserved tissue is sufficient for enrollment of the patient.
11. No treatment with biologic therapy, immunotherapy, chemotherapy, investigational agent for malignancy, or radiation ≤ 21 days before study registration.
12. No participation in another clinical trial in the period 30 days prior to start of first dose.
13. Patients should have resolution of any toxic effects of prior therapy (except alopecia) to NCI CTCAE, version 5.0, grade 1 or less.
14. Not pregnant and not nursing; for women of childbearing potential who are sexually active, a negative pregnancy test (urinary or serum beta-HCG) done ≤ 7 days prior to treatment start is required.
15. Absolute neutrophil count (ANC) ≥ 1,000/mm3.
16. Platelet count ≥ 70,000/mm3.
17. Creatinine ≤ 1.5 x upper limit of normal (ULN) OR calculated (calc.) creatinine clearance > 45 mL/min.
18. Total bilirubin ≤ 1,5 x upper limit of normal (ULN). If total bilirubin is greater than 1,5 x ULN, measure indirect bilirubin to evaluate for Gilbert's syndrome (if direct bilirubin is within normal range, participant may be eligible).
19. AST/ALT ≤ 2.5 x upper limit of normal (ULN).
20. Adequate pulmonary function (FEV1 > 2 liters or ≥ 75% of predicted for height and age).
21. No clinical significant heart failure (NYHA<III) or ejection fraction (echocardiography or scintigraphy; EF > 40%)
22. Female participants must be postmenopausal (no spontaneous menses for at least 2 years), surgically sterile (have had a hysterectomy or bilateral oophorectomy, tubal ligation, or otherwise be incapable of pregnancy), abstinent (at the discretion of the investigator), or if sexually active, have agreed to use an highly effective contraceptive method for the duration of their study participation (see Appendix 3 for guidance); patients should maintain adequate contraception for a minimum of 2 months after the last dose of dinutuximab beta. Male participants must agree to use an adequate contraception method as deemed appropriate by the investigator (e.g., vasectomy, double-barrier, partner using effective contraception) and to not donate sperm for a minimum of 5 months after treatment discontinuation.

Exclusion Criteria:

1. Symptomatic, untreated, or uncontrolled brain metastases present.
2. Patients with a known history of hypersensitivity to interleukin-2.
3. Patients with a hypersensitivity to zoledronic acid or to other bisphosphonates.
4. Need for invasive dental procedures. Preventive dental exams should be performed before starting zoledronic acid.
5. Patients after allogenic stem cell transplantation or other allogenic organ transplantation (e.g., liver, kidney etc.).
6. Patients with different malignant diseases other than sarcoma (measurable manifestations in the last 12 months or active therapy against the other malignant disease in the last 12 months).
7. Known active pulmonary disease with hypoxia defined as:

   * Oxygen saturation < 85% on room air or
   * Oxygen saturation < 88% despite supplemental oxygen.
8. Uncontrolled intercurrent illness including, but not limited to, poorly controlled hypertension or diabetes, ongoing active infection, or psychiatric illness/social situation that may potentially impair the participant's compliance with study procedures.
9. Patients who have received prior anti-GD2 therapy, including chimeric antigen receptor (CAR) T cells directed against GD2 antigen.
10. Lactating females are not eligible unless they have agreed not to breastfeed their infants.
11. Any condition that, in the opinion of the investigator, would compromise the well-being of the participant or the study or prevent the participant from meeting or performing study requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to assess the feasibility of the combined treatment with dinutuximab beta, zoledronic acid and low-dose interleukin 2. | 3 years, at EOS
  Feasibility rate, defined as the number of patients still on treatment and progression-free at Cycle 4 Day 5 divided by the number of all treated subjects.

SECONDARY OUTCOMES:
A secondary objective of this study is to assess the safety and tolerability of the combined treatment with dinutuximab beta, zoledronic acid and low-dose interleukin 2. | 3 years, at EOS
  To assess the safety and tolerability of the combined treatment of dinutuximab beta, zoledronic acid and low-dose interleukin-2 in patients with leiomyosarcomas, all adverse events will be assessed, and any alteration to the protocol in relation to study treatment will be assessed (e.g. discontinuation, reduction or delay of the treatment including the reasons for alterations of the predefined study treatment schedule).
An additional secondary objective of this study is to assess the efficacy of the combined treatment with dinutuaseximab beta, zoledronic acid and low-dose interleukin 2. | 3 years, at EOS
  Progression-free Survival (PFS) and Progression-free Survival after 6 months (PFSR6)
An additional secondary objective of this study is to assess the efficacy of the combined treatment with dinutuaseximab beta, zoledronic acid and low-dose interleukin 2. | 3 years, at EOS
  Masurement of Overall Response Rate (ORR).
An additional secondary objective of this study is to assess the efficacy of the combined treatment with dinutuaseximab beta, zoledronic acid and low-dose interleukin 2. | 3 years, at EOS
  Measurement of Overall Survival (OS).

OTHER OUTCOMES:
Tertiary/exploratory objective of this study is to evaluate and compare GD-2 immuno-histochemistry staining on cryopreserved and paraffin-embedded sarcoma tissue samples for future assessment of patient eligibility for anti-GD-2 therapy. | 3 years, at EOS
  To evaluate the GD2 immuno-histochemistry staining on cryopreserved and paraffin-embedded sarcoma tissue samples to identify patients eligible for treatment with dinutuximab beta, the staining methods and scores of GD2 expression on the different tissues will be compared.

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - HELIOS Klinikum Bad Saarow, Bad Saarow
  - Helios Klinikum Berlin-Buch, Berlin

IPD SHARING:
Plan to Share IPD: No